CLINICAL TRIAL: NCT01519492
Title: A Phase 2, Open-Label, Multi-Center Study of Safety, Tolerability, and Efficacy of AFN-12520000 in the Treatment of Acute Bacterial Skin and Skin Structure Infections (ABSSSI) Due to Staphylococci
Brief Title: A Study of Safety, Tolerability, and Efficacy of AFN-12520000 in the Treatment of Acute Bacterial Skin and Skin Structure Infections Due to Staphylococci
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affinium Pharmaceuticals, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12520000-010
Record Dates: First submitted 2012-01-17; First posted 2012-01-27 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections; Wound Infection; Cutaneous Abscess; Burn Infection; Cellulitis
Keywords: Skin and Subcutaneous Tissue Bacterial Infections
MeSH Terms: conditions — Wound Infection; Cellulitis | interventions — API 1252

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AFN-12520000 (Experimental): 100 mg tablet
  Interventions: Drug: AFN-12520000

INTERVENTIONS:
Drug: AFN-12520000 — Two tablets taken in both the morning and evening on an empty stomach for a total daily dose 400 mg
  Other Names: AFN-1252; API-1252

SUMMARY:
The purpose of the study is to determine the safety, tolerability and effectiveness of AFN-12520000 for in the treatment of Staphylococcal infections of the skin.

DETAILED DESCRIPTION:
This open-label Phase 2 study is designed as a proof-of-concept study to evaluate the efficacy of a total daily dose of 400 mg of AFN-12520000 using a number of newly defined early endpoints, conventional endpoints, and composite endpoints to determine clinical response. Safety and tolerability will also be evaluated by conventional endpoints.

The study will enroll up to 100 patients with a clinically documented diagnosis of Acute Bacterial Skin and Skin Structure Infections (ABSSSI) due to staphylococci. Patients meeting eligibility criteria will be identified and evaluated in a hospital or specialized clinic. After consent is obtained, the first dose of study medication will be administered. Daily clinical assessments will be conducted at the hospital and/or outpatient clinic during the first 5 days of treatment. Adverse events (AEs) and response to therapy will also be assessed.

The study will consist of a screening period, which includes the baseline visit; a treatment period, and an end-of-treatment (EOT) visit; and a follow-up period, which includes a short-term (Test-of-Cure [TOC]) follow-up (STFU/TOC) visit and a long-term follow-up (LTFU) visit.

Treatment regimens as short as 5 days (10 doses) and as long as 14 days (28 doses) will be permitted depending on individual response to treatment. The anticipated time commitment for patient participation in the study will be approximately 20 to 42 days from screening/baseline to the LTFU visit. The total duration of the study will be < 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and to understand the demands of the protocol;
* Ages of 18 and 70 years, inclusive;
* Have clinically documented ABSSSI suspected or documented to be caused by staphylococci accompanied by redness, edema, and/or induration of a minimum surface area of 75 cm2 and can be categorized as one or more of the following: Wound infection; Cutaneous abscess Burn infection (≤20% of total body surface area) or Cellulitis
* Have a primary infected lesion with at least three of the following: Significant pain or tenderness to palpation; Purulent or seropurulent drainage or discharge; Erythema; Fluctuance; Induration; Edema; Heat or localized warmth;
* Have at least two of the following signs and symptoms of systemic inflammation or complicating factors: Documented or reported fever >38.0°C; WBC count of >10,000 cells/mm3; Greater than 15% immature neutrophils irrespective of total WBC; Elevated CRP or ESR; or Local/regional lymphadenopathy;
* Have a Gram stain with Gram-positive cocci in clusters or PCR result indicating an infection with Staphylococci.
* Have clearly failed as defined in the protocol previous treatment after a minimum of 48 hours
* Women of childbearing potential must have a negative pregnancy test at screening before enrollment
* Male and Female patients must utilize a highly effective method of contraception
* In the judgment of the Investigator have an expectation of survival and prompt improvement with effective oral antibiotic therapy and appropriate supportive care for the anticipated duration of the study
* Willing and able to comply with all the study activities and procedures in the hospital or clinic.

Exclusion Criteria:

* Have any one of the following conditions:

  * Chronically infected "diabetic foot ulcers" or infections of chronic non-healing wounds of peripheral sites in a patient with advanced peripheral vascular disease;
  * A wound infection involving foreign body or prosthetic material that will not be removed within 48 hours of initiation of treatment;
  * Infected abdominal wounds unable to be surgically closed;
  * Necrotizing fasciitis, rapidly necrotizing infections, or gangrenous processes;
  * Infected burn involving >20% of the total body surface area;
  * Infected bite from human or animal origin.
  * Erysipelas or a primary infection suspected or documented to be due to streptococci or infection with a Gram-negative pathogen without evidence of a concomitant staphylococcal infection
  * Evidence of either a Gram-negative or Gram-positive pathogen not susceptible to treatment with protocol-specified antibiotics and AFN-12520000; or
  * An existing abscess that cannot be drained within 48 hours of initiation of treatment;
* Unable to tolerate an oral formulation of antibiotic, have an underlying gastrointestinal disease (would be poorly absorbed or tolerated), have a medical condition or post-operative condition leading to significant gastrointestinal malabsorption, and/or are unable to tolerate a normal diet;
* Have a known or suspected non-skin source of infection such as endocarditis, osteomyelitis, retroperitoneal abscess, septic arthritis, meningitis, or pneumonia;
* Exhibit signs of severe sepsis:
* Plans to have surgery utilizing general anesthetic during the study period (except surgery to remove a prosthetic device complicating the infection site or surgery to drain the abscess/wound within 48 hours);
* Pregnant or breastfeeding women;
* History of epilepsy, known seizure disorder, or history of severe and frequent migraine headaches;
* Taken an investigational medication during the month prior to enrollment;
* Prior exposure to the AFN investigational product;
* Known hypersensitivity to the protocol specified antibiotic necessary for the treatment of Staphylococcus or the protocol-specified concomitant antibiotic for the treatment of bacterial co-pathogens present in the wound;
* Treatment with any systemic antibiotic (excluding topical antibiotics), which is potentially effective against prevalent community or hospital isolates of Staphylococcus causing ABSSSI within 72 hours prior to enrollment and treatment with study medication unless the patient has clearly failed treatment;
* Not expected to survive for at least 60 days after enrollment;
* Anticipated amputation during the study of the limb involving the primary site of infection;
* History of human immunodeficiency virus infection with a current or previous CD4 count <200/mm3;
* Presence of immunodeficiency or an immunocompromised condition including hematologic malignancy, bone marrow transplant, or receiving immunosuppressive therapy such as cancer chemotherapy, medications for the rejection of transplantation, and long-term (≥2 weeks) use of systemic corticosteroids;
* Neutropenia
* End-stage renal disease or significant hepatic insufficiency
* Need for protocol defined prohibited concomitant treatments
* Unable or unwilling, in the judgment of the Investigator, to comply with the protocol
* An employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety | From time of consent to long term follow-up (max of 42 days)
  To assess the safety, tolerability, and efficacy of AFN-12520000 in patients with staphylococcal ABSSSI by exploring a variety of endpoints of clinical response and the rate and type of adverse events from baseline to the long term follow-up.

SECONDARY OUTCOMES:
Pharmacokinetics | Day 3, Day 5 and at EOT
  To assess the population pharmacokinetics (PK) of AFN 12520000 in patients with staphylococcal ABSSSI. PK measures will include Area Under the Curve (AUC), Maximum concentration (Cmax) and Half-life.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Hafkin, MD, Study Director — Affinium Pharmaceuticals, Ltd
Locations (14):
- United States (12):
  - SITE 018, Buena Park, California
  - SITE 005, Chula Vista, California
  - SITE 001, La Mesa, California
  - SITE 016, Oceanside, California
  - SITE 017, Augusta, Georgia
  - SITE 002, Columbus, Georgia
  - SITE 004, Savannah, Georgia
  - SITE 006, Las Vegas, Nevada
  - SITE 003, Somers Point, New Jersey
  - SITE 007, Cincinnati, Ohio
  - SITE 011, Toledo, Ohio
  - SITE 008, Nashville, Tennessee
- Canada (2):
  - SITE 014, Edmonton, Alberta
  - SITE 015, Kingston, Ontario

REFERENCES:
- [Derived] Hafkin B, Kaplan N, Murphy B. Efficacy and Safety of AFN-1252, the First Staphylococcus-Specific Antibacterial Agent, in the Treatment of Acute Bacterial Skin and Skin Structure Infections, Including Those in Patients with Significant Comorbidities. Antimicrob Agents Chemother. 2015 Dec 28;60(3):1695-701. doi: 10.1128/AAC.01741-15. PMID 26711777